CLINICAL TRIAL: NCT04383184
Title: Relationship Between Tracheal and Left Pulmonary Artery Stenosis Index and Prognosis of Pulmonary Artery Sling With Tracheal Stenosis
Brief Title: Relationship Between Tracheal and Left Pulmonary Artery Stenosis Index and Prognosis of PA Sling With Tracheal Stenosis
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020(40)
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Anomalies of Pulmonary Artery, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TRACHEAL FORMING GROUP: Left pulmonary artery transplantation and slide tracheoplasty
  Interventions: Procedure: tracheoplasty
- NON-TRACHEAL FORMING GROUP: only Left pulmonary artery transplantation
  Interventions: Procedure: tracheoplasty

INTERVENTIONS:
Procedure: tracheoplasty — tracheoplasty and only left pulmonary artery transplantation

SUMMARY:
Pulmonary artery sling is a rare congenital pulmonary vascular malformation, often associated with tracheal or bronchial stenosis. Surgical treatment of pulmonary artery sling with tracheal stenosis has a high risk and a relatively poor prognosis. This article aims to explore the relationship between the index of tracheal and left pulmonary artery stenosis and the surgical effect of pulmonary artery sling with tracheal stenosis. Methods: Retrospective analysis of the cases of pulmonary artery sling surgery in our center from January 2010 to December 2018. Before operation, routine cardiac enhancement CT examination was performed, and the diameter of the left pulmonary artery and the tracheal stenosis were measured on the CT tomogram respectively, and the ratio of the degree of tracheal stenosis / left pulmonary artery stenosis (T / P) was calculated, combining the surgical method and clinical prognosis analyzed and discussed.

DETAILED DESCRIPTION:
Pulmonary artery sling is a rare congenital pulmonary vascular malformation. The abnormality of the left pulmonary artery originates from the right pulmonary artery instead of the trunk of the pulmonary artery. It passes around the trachea, passes between the trachea and the esophagus, and forms a vascular ring with the arterial ligament. Compression of the trachea and esophagus, especially the symptoms of tracheal stenosis caused by the compression of the trachea, can be manifested as serious symptoms such as respiratory infections, wheezing, and even respiratory distress, which can be life-threatening in severe cases. Therefore, the key to the surgical treatment of pulmonary artery sling is to relieve tracheal compression and correct tracheal stenosis, which is also the difficulty. At present, the overall survival rate of surgical treatment of pulmonary artery sling around the world is about 78% to 93% [1], but the mortality rate for patients with severe tracheal stenosis is also high, reaching about 24% [1], mainly due to pre-operative or post-operative respiratory failure caused by narrowed trachea. At present, the selection and intervention of pulmonary artery sling combined with tracheal stenosis is still a difficult problem. On the one hand, if tracheoplasty is performed, anastomotic scar hyperplasia after surgery may lead to local tracheal stenosis again [2], and long-term care is also quite difficult; If tracheoplasty is not performed, tracheal stenosis may not be completely relieved, and obstructive ventilation disorder and respiratory failure may occur after surgery [1]. At present, there is basically no objection to the preoperative assessment methods of pulmonary artery sling. CCTA is generally considered to be an effective method for diagnosing pulmonary artery sling with tracheal stenosis. It can display abnormally deformed pulmonary arteries and narrowed trachea, and it can also detect intracardiac malformations. The important means of preoperative evaluation can also be used for postoperative evaluation [3].

There is currently no consensus on the indications for tracheal intervention with pulmonary artery sling combined with tracheal stenosis. Some researchers believe that tracheoplasty should be performed for tracheal diameters less than 3mm, or the prognosis is poor [4]. Some researchers have suggested that the diameter / length percentage of tracheal stenosis can be used as a reference index for intervention of tracheal stenosis [5]. Brouns et al. found that the square of the cross-sectional area of the tracheal stenosis has a significant proportional relationship with the air flow, so they believe that the cross-sectional area of the tracheal stenosis is the main factor affecting the ventilation effect [6]. When I reviewed the imaging data of children with tracheal stenosis in our center, the most severe tracheal stenosis is usually located in the vascular ring formed by the right pulmonary artery starting segment, the left pulmonary artery starting segment, and the left pulmonary artery bypass segment. Not only was the trachea compressed and significantly narrowed, but the left pulmonary artery was also significantly narrowed, that is, the trachea and the left pulmonary artery were squeezed together in a limited space, causing both of them to be compressed and narrowed. This study was the first to investigate the interaction and morphological changes of the trachea and the left pulmonary artery, and the ratio of the degree of tracheal stenosis / left pulmonary artery stenosis (T / P) was used to indicate the degree of interaction between the two. A larger T / P ratio indicates that the left pulmonary artery is more dominant in tracheal compression, and tracheal stenosis is usually more serious. On the contrary, a smaller T / P ratio indicates that the trachea is more dominant in compression of the left pulmonary artery, and the tracheal stenosis is usually relatively lighter. This article retrospectively analyzes the cases in our center and discusses the effects of surgical treatment.

ELIGIBILITY:
Inclusion Criteria: surgical cases of pulmonary artery sling operated in our center from January 2010 to December 2018 -

Exclusion Criteria:cases of pulmonary artery sling without opertion

-

Ages: 1 Month to 57 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with tracheoplasty and left pulmonary artery transplantation at the same time, and only with left pulmonary artery transplantation
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of tracheal forming group and non-tracheal forming group | 30 days
  Tracheal stenosis (T) and left pulmonary artery stenosis (P) ratio were compared between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No